CLINICAL TRIAL: NCT04117542
Title: Neural Substrates of Context-dependent Working Memory in Youth With Overweight/Obesity and Loss of Control Eating
Brief Title: Working Memory in Overweight Children With and Without Loss of Control Eating
Status: Completed | Type: Observational
Sponsor: The Miriam Hospital (Other)
Collaborators: Brown University (Other)
Responsible Party: Sponsor
Other Study IDs: 1205595
Record Dates: First submitted 2019-10-02; First posted 2019-10-07 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2019-10

CONDITIONS: Binge Eating; Pediatric Obesity
Keywords: Loss of Control Eating; Working Memory
MeSH Terms: conditions — Bulimia; Pediatric Obesity | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Overweight/Obesity Control: Adolescents who have overweight/obesity, but do not report loss of control eating.
  Interventions: Other: Observational
- Overweight/Obesity Experimental: Adolescents who have overweight/obesity, and report loss of control eating.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational data will be obtained through participant self-response, parental response, cognitive performance, and neural imaging.

SUMMARY:
Loss of control (LOC) eating in children is associated with multiple physical and mental health impairments, including obesity and eating disorders. Little is known about the developmental neurobiology of LOC, which is crucial to specifying its pathophysiology and the development of effective preventive interventions. Individual differences in working memory (WM) appear to be related to LOC eating and excess weight status in youth, but the specificity and neural correlates of these individual differences are unclear. Failure to adequately understand the nature of associations between WM and eating behavior in children with overweight/obesity limits the development of appropriately-targeted, neuro-developmentally informed interventions addressing problematic eating and related weight gain in youth. To close this clinical research gap, the current study proposes to investigate the context-dependence of WM impairment and its neural correlates in children with concomitant overweight/ obesity and LOC eating as compared to their overweight/obese peers.

Specific aims are to investigate:

1)WM performance in youth with LOC eating relative to overweight/obese controls during recalls in the context of food-related versus neutral distractors; and 2) neural activation patterns during WM performance across both food-related and neutral stimuli. We hypothesize that, relative to their overweight/obese peers, youth with LOC eating will show 1) more errors and slower response times during recalls involving food-related vs. neutral distractors, and fewer errors and faster response times during recalls involving food-related vs. neutral targets; 2) increased activation in prefrontal regions during WM performance across stimuli types relative to overweight/obese controls, and 3) even greater activation in the context of food-related versus neutral distractors.

The proposed study is the first to use state-of-the-science neuroimaging methodology to clarify the relations between WM and LOC eating, with strong potential to advance understanding of the associations among executive functioning, excess weight status, and eating pathology, and inform the development of interventions (e.g., WM training) to alleviate their cumulative personal and societal burden.

ELIGIBILITY:
Inclusion Criteria:

* Overweight/Obese (>85% expected body mass)
* Right-handed

Exclusion Criteria:

* Currently taking any medications known to affect their weight/appetite
* Report current or past medical or psychiatric conditions known to significantly affect eating or weight (e.g., diabetes, bulimia nervosa), with the exception of binge eating disorder
* Have an intelligence quotient (IQ) in the borderline range or lower, or any condition affecting executive functioning (e.g., recent concussion, history of traumatic brain injury)
* Are unable to read or comprehend study materials
* Are receiving concurrent treatment for overweight/obesity
* Have metallic foreign bodies, face or neck tattoos, or other conditions that would prohibit fMRI scanning

Ages: 10 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Participants will be 30 children, ages 10-17, 15 of whom who are overweight/obese and report loss of control eating (i.e., at least 3 objectively or subjectively large loss of control episodes in the past 3 months), and 15 of whom who will serve as overweight/obese controls.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
BMI | 1 day
  Body Mass Index calculated with height/weight (cm/g)
Eating Behavior | 1 day
  Eating behavior will be assessed using the Eating Disorders Examination (EDE), a semi-structured interview.
Neural Activity | Up to 2 weeks
  Neural activation will be assessed using functional magnetic resonance imaging (fMRI) data
Working Memory | 1 day
  Working memory will be assessed using the NIH Toolbox list sort task.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea B. Goldschmidt, Ph.D., Principal Investigator — Warren Alpert Medical School of Brown University
Locations (1):
- Weight Control & Diabetes Research Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/42/NCT04117542/ICF_000.pdf